CLINICAL TRIAL: NCT05688696
Title: A Phase IIb, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients With Systemic Lupus Erythematosus
Brief Title: Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICP-CL-00124
Record Dates: First submitted 2023-01-10; First posted 2023-01-18 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Systemic Lupus Erythematosus, SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orelabrutinib Lower Dose (Experimental)
  Interventions: Drug: Orelabrutinib (Low Dose)
- Orelabrutinib Higher Dose (Experimental)
  Interventions: Drug: Orelabrutinib (High Dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Orelabrutinib Placebo

INTERVENTIONS:
Drug: Orelabrutinib (Low Dose) — Subjects will be administered with lower dose of Orelabrutinib orally once daily in combination with SOC therapy
  Arms: Orelabrutinib Lower Dose
Drug: Orelabrutinib (High Dose) — Subjects will be administered with higher dose of Orelabrutinib orally once daily in combination with SOC therapy
  Arms: Orelabrutinib Higher Dose
Drug: Orelabrutinib Placebo — Subjects will be administered with Orelabrutinib Placebo orally once daily in combination with SOC therapy
  Arms: Placebo

SUMMARY:
This is a phase IIb, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of orelabrutinib in adult subjects with SLE who are receiving standard of care (SOC) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. have had a detailed understanding of the nature, significance, potential benefits, potential risks, and procedures of the study, and voluntarily signed a written Informed Consent Form (ICF).
2. Males or females aged≥18 and ≤75 years.
3. Have a clinical diagnosis of SLE 6 months prior to signing the ICF, meeting at least 4 of the 11 American College of Rheumatology (ACR) classification criteria for SLE.
4. SLEDAI-2K≥8 at screening.
5. Are on a stable SLE SOC therapy consisting of any of the following medications for a period of at least 30 days prior to the first dose: glucocorticoid, and/or anti-malarials, and/or immunosuppressive agents.
6. Have a positive test for anti-dsDNA antibody (> normal range) and/or anti-nuclear antibody (ANA) and/or anti-Smith antibody at screening.
7. Women of childbearing potential must take a complementary barrier method of contraception in combination with a highly effective method of contraception at screening, throughout the trial, and within 90 days after the last dose of the investigational agent. In this trial.

Exclusion Criteria:

Medical conditions:

1. Pregnant or lactating women, and men or women who have birth plans in the past 12 months.
2. Have neuropsychiatric systemic lupus erythematosus (NPSLE) within 6 months prior to the first dose, including seizures, psychosis, organic brain syndrome, cerebrovascular accident, cranial neuropathy, cerebritis, cerebral vasculitis or lupus headache.
3. Have severe lupus nephritis, or have required hemodialysis or high-dose glucocorticoid within 90 days prior to the first dose.
4. Have autoimmune diseases other than SLE (excluding secondary Sjogren's syndrome).
5. Have a history of any non-SLE disease that has required treatment with oral or intravenous or intramuscular or subcutaneous injection glucocorticoids for more than a total of 2 weeks within the last 24 weeks prior to signing the ICF.
6. Have a history of or current diagnosis of Central Nervous System (CNS) diseases.
7. Have clinically documented cardiovascular diseases that are obviously unstable or not effectively treated.
8. Have significant active lung diseases (e.g., interstitial lung disease, obstructive pulmonary disease).
9. Have severe hepatobiliary diseases.
10. Have a history of malignant neoplasm.
11. Have a history of a major organ transplant or hematopoietic stem cell/marrow transplant.
12. Have known allergies to any component of the investigational agent as described in the Protocol.

    Concomitant medication and surgery:
13. Have received rituximab, epratuzumab, or any other B cell-depleting therapy within 12 months prior to randomization.
14. Have received cyclophosphamide and chlorambucil within 6 months prior to randomization.
15. Have received belimumab, tumor necrosis factor (TNF) blockers, interleukin receptor blockers or other biological agents within 3 months prior to randomization (or 5 half-lives, whichever is longer).

    Lab tests:
16. Have a positive test for human immunodeficiency virus (HIV) antibody.
17. Have a positive test for Hepatitis B Surface Antigen (HBsAg) or hepatitis C antibody, or have a positive test for hepatitis B virus (HBV) DNA by Polymerase Chain Reaction (PCR) if positive for Hepatitis B Core Antibody (HBcAb).
18. Have abnormal tissue or organ function, meeting any of the following at screening:

    * Absolute neutrophil count (ANC) < 1.5 × 10^9/L; hemoglobin < 90 g/L; lymphocyte count < 0.8 × 10^9 /L.
    * Calculated estimated glomerular filtration rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation < 45 mL/min/1.73 m2.

    Others:
19. Have other conditions that are not appropriate for participation in the trial as considered by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
SLE Responder Index (SRI) - 4 response rate | Week 48
  SRI-4 response is defined as: 1)≥4 point reduction from baseline in SLE disease activity index-2000 (SLEDAI-2K) score; 2) no worsening (increase of <0.3 points from baseline) in Physician's Global Assessment (PGA); 3) no new A organ domain score or no more than 1 new B organ domain scores compared with baseline in British Isles Lupus Assessment Group (BILAG)-2004.

SECONDARY OUTCOMES:
SLE Responder Index (SRI) - 6 response rate | Week 48
  SRI-6 response is defined as: 1)≥6 point reduction from baseline in SLE disease activity index-2000 (SLEDAI-2K) score; 2) no worsening (increase of <0.3 points from baseline) in Physician's Global Assessment (PGA); 3) no new A organ domain score or no more than 1 new B organ domain scores compared with baseline in British Isles Lupus Assessment Group (BILAG)-2004.
British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) response rate | Week 48
  BICLA response is defined as: 1) In BILAG-2004, reduction of all baseline A to B/C/D and baseline B to C/D, and no worsening in other organ systems (as defined by no new A organ domain score or no more than 1 new B organ domain scores); 2) No worsening from baseline in SLEDAI-2K, where worsening is defined as an increase from baseline of >0 points in SLEDAI-2K; 3) No worsening (increase of <0.3 points from baseline) in PGA.
Time to 1st flare | Week 48
The proportion of subjects whose average prednisone dose has been reduced by≥25% from baseline to ≤7.5 mg/day | Week 48
Changes from baseline in the levels of complement C3, complement C4, and anti-dsDNA antibody | Week 48
  Adopt the unified unit standard of central laboratory testing
Treatment Emergent Adverse Events, Treatment Related Adverse Events, Treatment Emergent Serious Adverse Events, Treatment Related Serious Adverse Events. | Up to Week 52
Mean change from baseline in the 36-Item Short Form Health Survey (SF-36) scores (The SF-36 consists of eight domains. Each domain score ranges from 0-100. The higher the score, the better the health. ) | Week 48

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of XiaMen University, Xiamen, Fujian
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - The first affiliated hospital of shantou university medical college, Shantou, Guangdong
  - The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Affiliated Hospital of HeBei University, Baoding, Hebei
  - Hebei People's Hospital, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The first hospital of Qiqihar, Qiqihar, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second XIANGYA Hospital Of Central South University, Changsha, Hunan
  - Yiyang Central Hospital, Yiyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiujiang NO.1 People's Hospital, Jiujiang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - Shengjing Hospital of china medical university, Shenyang, Liaoning
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Nei Monggol Autonomous Region
  - Affiliated Hospital of Binzhou Medical College, Binzhou, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - The Third People's Hospital of Huzhou, Huzhou, Zhejiang
  - The First Hospital of Ningbo, Ningbo, Zhejiang
  - The First People's Hospital of Wenling, Wenling, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No